CLINICAL TRIAL: NCT03737227
Title: Analysis of Lumbar Intervertebral Motion During Flexion and Extension Cinematographic Recordings in Asymptomatic Male Participants.
Brief Title: Lumbar Intervertebral Motion in Asymptomatic Male Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL63033.096.18
Record Dates: First submitted 2018-11-02; First posted 2018-11-09 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-02

CONDITIONS: Lumbar Intervertebral Motion
Keywords: Lumbar intervertebral motion; Flexion; Extension; Cinematographic recording; Segmental rotations; Segmental translation; lumbar spine; asymptomatic participants

STUDY DESIGN:
Intervention Model Description: Fundamental research with 11 male participants in one study arm, all performingflexion and extension of the lumbar spine during cinematographic recordings twice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cinematographic recording (Other): Cinematographic recordings of the asymptomatic participants during flexion and extension of the lumbar spine.Cinematographic recordings will be performed twice with an interval of two weeks.
  Interventions: Radiation: Cinematographic recording

INTERVENTIONS:
Radiation: Cinematographic recording — Cinematographic recording during flexion and extension of the lumbar spine.

SUMMARY:
The investigators aim to analyze the physiological segmental motion of the lumbar spine during flexion and extension cinematographic recordings of asymptomatic individuals.

DETAILED DESCRIPTION:
In this study the investigators aim to define the lumbar spines' physiological motion by analyzing sequence of initiation of motion and sequence of maximum contribution in segmental translation and rotation of each vertebra L1, L2, L3, L4, L5 and S1 by using flexion and extension cinematographic recordings in asymptomatic male participants. Participants will undergo two cinematographic recordings with an interval of two weeks. Segmental translation and rotation of each segment will be plotted against total range of motion of the lumbar spine for each individual participant. With these graphs the investigators can analyze if there are specific physiological motion patterns during flexion and extension of the lumbar spine. In the future, the investigators hope to compare these physiological motion patterns to potential abnormal motion patterns in patients suffering from lumbar spinal pathology or after lumbar spine surgery to gain knowledge about complaints and, for example, adjacent level disease.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 18 and 25 years old.
* BMI under 25
* Participants have to be able to perform flexion and extension over a full range of motion without complaints of pain.
* Participants have no medical history of spinal problems based on anamneses and zero ODI-, and VAS-score.
* Kellgrens' classification on cinematographic recordings is zero or one.
* Informed consent has been signed.
* Ability to read and understand Dutch.

Exclusion Criteria:

* Medical history of visiting general practitioners, allied health professionals or specialists for spinal problems.
* Former spine surgery.
* Radiographs of abdomen, pelvis, hips, lumbar spine or sacral spine in last year.
* Degenerative abnormalities of the lumbar spine.
* Active spinal infection.
* Immature bone.
* Lumbar tumor processes.
* Former lumbar radiotherapy.
* Congenital lumbar spine abnormalities, for example spina bifida.
* Planning pregnancy for the coming year.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Lumbar segmental rotation | 30 minutes
  Analyzing sequence of initiation of motion and sequence of segmental contribution in rotation of each vertebra L1, L2, L3, L4, L5 and S1 by using flexion and extension cinematographic recordings in asymptomatic male participants.

SECONDARY OUTCOMES:
Lumbar segmental translation | 30 minutes
  Analyzing intervertebral horizontal and vertical translation of each vertebra L1, L2, L3, L4, L5 and S1 by using flexion and extension cinematographic recordings in asymptomatic male participants. If mean intra-class correlation coefficient is higher than 0.60, sequence of initiation of motion and sequence of segmental contribution of intervertebral horizontal and vertical translation will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Henk Van Santbrink, Dr., Principal Investigator — neurosurgeon Zuyderland
Locations (1):
- Zuyderland Medical Center, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caelers I, Boselie T, van Hemert W, Rijkers K, De Bie R, van Santbrink H. The Variability of Lumbar Sequential Motion Patterns: Observational Study. JMIR Biomed Eng. 2023 Jun 20;8:e41906. doi: 10.2196/41906. PMID 38875682
- [Derived] Caelers IJ, Boselie TF, Rijkers K, Van Hemert WL, De Bie RA, Van Santbrink H. Lumbar Intervertebral Motion Analysis During Flexion and Extension Cinematographic Recordings in Healthy Male Participants: Protocol. JMIR Res Protoc. 2020 Feb 24;9(2):e14741. doi: 10.2196/14741. PMID 32130199

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT03737227/Prot_SAP_000.pdf